CLINICAL TRIAL: NCT06240169
Title: Effect of Age on the Success of Direct Pulp Capping Using Bio-ceramic Materials in Cariously Exposed Teeth With Reversible Pulpitis: A Prospective Clinical Study.
Brief Title: Effect of Age on the Success of DPC Using Bio-ceramic Materials in Cariously Exposed Teeth With Reversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Harshita Wadhwa
Record Dates: First submitted 2024-01-14; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Pulpitis Reversible
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the outcome assessors will be blinded to the allocation groups (double-blinding). But the operator (Principal investigator) will not be blinded due to the nature of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- DPC in AGE I with MTA (Experimental): DPC using MTA in Age group I i.e. 18-40years.
  Interventions: Procedure: DPC with MTA in AGEI
- DPC in AGE I with BD (Experimental): DPC using BD in Age group I i.e. 18-40years.
  Interventions: Procedure: DPC with BD in AGEI
- DPC in AGE II with MTA (Experimental): DPC using MTA in Age group II i.e. 41-60years
  Interventions: Procedure: DPC with MTA in AGEII
- DPC in AGE II with BD (Experimental): DPC using BD in Age group II i.e. 41-60years
  Interventions: Procedure: DPC with BD in AGEII

INTERVENTIONS:
Procedure: DPC with MTA in AGEI — DPC using MTA in 18-40 years
  Arms: DPC in AGE I with MTA
Procedure: DPC with BD in AGEI — DPC using BD in 18-40 years
  Arms: DPC in AGE I with BD
Procedure: DPC with MTA in AGEII — DPC using MTA in 41-60Years
  Arms: DPC in AGE II with MTA
Procedure: DPC with BD in AGEII — DPC using BD in 41-60Years
  Arms: DPC in AGE II with BD

SUMMARY:
Study Title: - Effect of age on the success of direct pulp capping using bio-ceramic materials in cariously exposed teeth with reversible pulpitis: A Prospective clinical study.

Rationale: - Preservation of pulp vitality is a critical factor in long-term tooth survival. In deep carious lesion with reversible pulpitis, vital pulp therapy procedures in the form of direct pulp capping(DPC)is more conservative treatment strategy, based on the premise that a biologically active material placed in direct contact with the pulp wound can determine the pulpal response and result in the development of a reparative hard tissue bridge to preserve pulp vitality. Patient's age may have a role in the survival rate after direct pulp capping and the role of the pulp capping material has been recognized as an important parameter for the success of treatment.

Research Question : Does age has any influence on the success of DPC procedure and is there any difference between MTA and Biodentine as DPC material in cariously exposed permanent teeth with reversible pulpitis? Aim & Objectives- To evaluate the effect of age on success of Direct Pulp Capping, to evaluate the success of MTA and Biodentine as direct pulp capping agents.

DETAILED DESCRIPTION:
Study Title: - Effect of age on the success of direct pulp capping using bio-ceramic materials in cariously exposed teeth with reversible pulpitis: A Prospective clinical study.

Rationale: - Preservation of pulp vitality is a critical factor in long-term tooth survival. In deep carious lesion with reversible pulpitis, vital pulp therapy procedures in the form of direct pulp capping(DPC)is more conservative treatment strategy, based on the premise that a biologically active material placed in direct contact with the pulp wound can determine the pulpal response and result in the development of a reparative hard tissue bridge to preserve pulp vitality. Patient's age may have a role in the survival rate after direct pulp capping and the role of the pulp capping material has been recognized as an important parameter for the success of treatment.

Research Question : Does age has any influence on the success of DPC procedure and is there any difference between MTA and Biodentine as DPC material in cariously exposed permanent teeth with reversible pulpitis? Aim & Objectives- To evaluate the effect of age on success of Direct Pulp Capping, to evaluate the success of MTA and Biodentine as direct pulp capping agents based on clinical and radiographic findings and assessment of post operative pain for 7 days post treatment.

Statistical method: - Data analysis by suitable statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA I and ASA II).
* Patients falling in the age group of 18-60 years.
* Restorable permanent mandibular posterior teeth.
* Extremely deep caries penetrating the entire thickness of dentine and exhibiting signs and symptoms of reversible pulpitis.
* Teeth responding positively to cold test and electric pulp testing with no tenderness on percussion.

Exclusion Criteria:

* Primary teeth.
* Traumatic or mechanical exposure.
* No pulp exposure after caries excavation.
* Hemostasis not achieved within 10 mins.
* Teeth with irreversible pulpitis.
* Presence of periapical lesion or evidence of internal or external resorption, calcified canals, as assessed by radiographic examination.
* Patients with periodontal disease, swelling and sinus tract.
* Immunocompromised or pregnant patients, patients with any systemic disease, and a positive history of antibiotic use within 1 month and analgesic use within week before the treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
clinical and radiographic success rates and evaluation of the effect of age on the success of procedure. | Baseline to 18 months
  CLINICAL SUCCESS CRITERIA
  * Absence of sign and symptoms of pain on stimulus or spontaneous pain.
  * Absence of tenderness to palpation or percussion and presence of functional tooth.
  * Absence of any soft tissue swelling sinus or fistula.
  * Normal tooth mobility and no periodontal probing depth.
  * Positive response to pulp sensibility test (cold and EPT).
  RADIOGRAPHIC SUCCESS CRITERIA
  * Periapical Index (PAI) score ≤2.
  * Absence of external or internal root resorption.
  Also, to evaluate the effect of age on the success of procedure.

SECONDARY OUTCOMES:
Post operative pain Secondary outcome measure will be pain intensity after treatment. Secondary outcome measure will be pain intensity after treatment. Secondary outcome measure will be pain intensity after treatment. | Base line to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Tewari, Principal Investigator — pgids rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No